CLINICAL TRIAL: NCT04944394
Title: Psychological and Ethical Support for Hospital Professionals During the COVID-19 Pandemic: Suitability and Post-crisis Implications for the Experience of All Professionals
Acronym: PsyCOVID All P
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: QUENOT 2020-3
Record Dates: First submitted 2021-06-28; First posted 2021-06-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Psychological Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospital professionals: all professionals working in hospitals in France
  Interventions: Other: online questionnaire; Other: questionnaire survey

INTERVENTIONS:
Other: online questionnaire — Administration of an online questionnaire (Limesurvey platform) at M0
  - This questionnaire includes a characterization of the professional (center, profession, usual department and department during the health crisis, family situation). Generic stress factors, the traumatic impact of the crisis and collective and individual coping strategies are also collected.
Other: questionnaire survey — A questionnaire survey of the chief physician of the intensive care unit of each hospital will make it possible to characterize the support provided by the institution and how it changed over time

SUMMARY:
SARS-COV-2 has created an unprecedented health crisis, resulting in unprecedented mobilization of all hospital professionals. The massive influx of patients overwhelmed the human, therapeutic and material resources available, and teams were confronted with an unusually heavy workload in a highly stressful emergency context. These professionals were thus exposed to a risk of over-investment in a context of acute and repetitive stress over an indefinite period of time, combining a heavy workload, emotional challenges and specific ethical issues. These factors simultaneously affected the professional sphere but also the personal and family spheres (lockdown, risk of contamination). In this context, the mental health of hospital staff is considered to be more important than ever, as emphasized on numerous occasions by the Director General of Health and the French Minister for Health and Solidarity. Mental health involves the way in which individuals respond specifically to work-related suffering by developing individual and collective defensive strategies. Thus, the question of the mental health of hospital professionals cannot be considered without taking into account the strategies implmented to combat stress, and the factors that contribute or not to the construction and stabilization of the work environment (collaboration, support).

ELIGIBILITY:
Inclusion Criteria:

All professionals working in hospitals Professionals involved in the organization of psychological and ethical support may also be interviewed to provide the information necessary to describe and evaluate the support provided and how it changed over time.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all professionals working in hospitals
Sampling Method: Non-Probability Sample
Enrollment: 4522 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Score assessed by Global Health Questionnaire GHQ-12 | at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Fournier A, Laurent A, Lheureux F, Ribeiro-Marthoud MA, Ecarnot F, Binquet C, Quenot JP. Impact of the COVID-19 pandemic on the mental health of professionals in 77 hospitals in France. PLoS One. 2022 Feb 16;17(2):e0263666. doi: 10.1371/journal.pone.0263666. eCollection 2022. PMID 35171915
- [Derived] Fournier A, Deltour V, Lheureux F, Poujol AL, Ecarnot F, Binquet C, Quenot JP, Laurent A. Association between burnout and PTSD, and perceived stress in the workplace among healthcare workers in the intensive care unit: a PsyCOVID-ICU substudy. Psychol Health Med. 2025 Apr;30(4):752-769. doi: 10.1080/13548506.2025.2454038. Epub 2025 Feb 10. PMID 39927681